CLINICAL TRIAL: NCT06922981
Title: Comparison Between Periodized Resistance and Aerobic Training Programs on Nonspecific Chronic Low Back Pain
Brief Title: Periodized Resistance and Aerobic Training in Non-Specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Saied mohammed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: periodized RT and AT in NSCLBP
Record Dates: First submitted 2023-12-22; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistance group (Experimental): Nineteen male and female patients aged 18 to 45 years, diagnosed with NSCLBP were recruited through referrals from orthopedic surgeons.The exercise program included upper and lower body resistance training exercises including leg press, lateral pull down, abdominal crunch, Swiss ball abdominal crunch, and prone superman exercises, utilizing free weights, machines, and bodyweight exercises. The therapist performed a one-repetition maximum (1 RM) test at baseline to determine the initial exercise loads. Participants then performed exercises at 50% to 70% of their 1 RM value. This process of periodic 1 RM testing and training at 50% to 70% of the value is repeated every two weeks till the end of the study.
  Interventions: Behavioral: resistance training program
- aerobic group (Experimental): Nineteen male and female patients aged 18 to 45 years, diagnosed with NSCLBP were recruited through referrals from orthopedic surgeons.The periodized aerobic training (AT) program consisted of three sessions per week. Each Exercise session consisted of a 5-minute warm-up, 30 minutes of aerobic exercise, and a 5-minute cool-down. Backward walking was performed on a motorized treadmill.The participants began with 10-15 minutes of exercise at 40-55% HRR (RPE=11-12, light) during the first two weeks, 20-30 minutes of exercise at 55-70% HRR (RPE=12-13, somewhat hard) during the third and fourth week, then 30 minutes of exercise at 70-85% HRR (RPE=14-16, hard) for the remainder of the study.
  Interventions: Behavioral: resistance training program

INTERVENTIONS:
Behavioral: resistance training program — Thirty-eight male and female patients aged 18-45 years, diagnosed with NSCLBP will be recruited through direct referrals from orthopedic surgeons, based on their availability to participate, thus a sample of convenience will be used, Participants will be randomly assigned as follows:
  Group A:
  Patients in group (A) (n=19) will receive a periodized resistance exercise program.
  Group B:
  The patients in group (B) (n=19) will receive a periodized aerobic exercise program
  Other Names: aerobic training program

SUMMARY:
The aim of the study is to compare the effectiveness of two forms of periodized exercise training programs (resistance and aerobic ) using the best recommended parameters (volume, intensity, rest period, and frequency) on the best available outcome measures (pain, disability, fear of movement, back and abdominal muscular endurance, upper body strength (latissimus dorsi muscle),and lower body strength ( gluteus maximus )

DETAILED DESCRIPTION:
Low back pain (LBP) is a significant health problem and the leading cause of disability throughout the world, representing one of the most common reasons for primary care physician visits, with a lifetime prevalence reported as high as about 80%. It causes a significant economic and social burden that will become even more daunting in the coming decades. People with LBP are 2.5 times more likely to experience psychological distress and pain compared to normal people, which can adversely affect quality of life. Low back pain is commonly classified as nonspecific or specific due to the reported cause and as acute (<6weeks), subacute (6-12 weeks), or chronic (>12weeks) according to the duration of symptoms. A periodized training model is considered more effective at improving the physiological function than non-periodized (basic progressive overload), as it allows progressive adjustment of volume and intensity of training program.periodization is defined as the planned manipulation of training variables (load, sets, and repetitions) in order to maximize training adaptations and to prevent the onset of overtraining syndrome. Various periodization models exist: undulating periodization comprises a frequent variation in stimuli between low, moderate, and high intensity typically on a weekly basis, whereas traditional linear periodization typically contains low load and high volume in the initial phase of training with a gradual shift towards high load and low volume as the training progresses. Periodization may also be beneficial due to adding variation to workouts by manipulating sets, repetitions, exercise order, number of exercises, resistance, rest periods, type of contractions, or training frequency. Another added benefit is the avoidance of training plateaus or boredom. Thus it seems reasonable to consider a periodized training model in the management of those with NSCLBP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with nonspecific (nonspecific pathology) chronic (> 12 weeks) low back pain (localized below the costal margin and above the gluteal fold) (Owen et al., 2020).

  * Participants aged between 18 to 45 years (Wewege et al., 2018).
  * Participants with Body Mass Index (BMI) 18.5-29.9 Kg/m2.
  * VAS score 3-8 cm (Pieler-Bruha, 2009).
  * ODI score 10-60 (Pieler-Bruha, 2009).

Exclusion Criteria:

* Participants will be excluded if they did not meet the inclusion criteria mentioned above such as pain due to or associated with:

  * Pregnancy
  * Infection
  * Fracture
  * Tumor
  * Structural deformity (e.g. scoliosis)
  * Radicular syndrome or cauda equine syndrome
  * Inflammatory disorders (Owen et al., 2020)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measured by Visual Analogue Scale (VAS) | baseline (week 0) and at the end of intervention (week 8)
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), a 10 cm horizontal scale where 0 cm represents "no pain" and 10 cm represents "worst imaginable pain." Participants will rate their pain at rest and during movement.
Disability Level Measured by the Oswestry Disability Index (ODI) | baseline (week 0) and at the end of intervention (week 8)
  Disability related to low back pain will be assessed using the Oswestry Disability Index (ODI), a validated 10-item questionnaire measuring limitations in daily activities due to pain. Each item is scored from 0 to 5, with total scores ranging from 0% (no disability) to 100% (severe disability). Higher scores indicate greater disability.
Fear of movement measured by Tampa Scale of Kinesiophobia (TSK) | baseline (week 0) and at the end of intervention (week 8)
  Fear of movement related to pain will be assessed using the Tampa Scale of Kinesiophobia (TSK), a validated 17-item questionnaire designed to measure fear of movement and injury-related avoidance behavior. Each item is scored on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree), with total scores ranging from 17 (low fear) to 68 (high fear).
Abdominal Muscular Endurance Measured by the Abdominal Muscular Endurance Test Abdominal Muscular Endurance Measured by the Abdominal Muscular Endurance Test Abdominal Muscular Endurance Measured by the Abdominal Muscular Endurance Test | baseline (week 0) and at the end of intervention (week 8)
  Abdominal endurance will be assessed using the Abdominal Muscular Endurance Test, which requires participants to perform a curl-up to the rhythm of a metronome for as long as possible.
Back Isometric Muscular Endurance Measured by the Biering-Sørensen Back Endurance Test Back Isometric Muscular Endurance Back Isometric Muscular Endurance Measured by the Biering-Sørensen Back Endurance Test (BSBE) | baseline (week 0) and at the end of intervention (week 8)
  Back endurance will be assessed using the Biering-Sørensen Back Endurance Test (BSBE), which evaluates the endurance of the lumbar extensor muscles. The test involves the participant holding a prone position on a plinth with the upper body suspended and supported only by the pelvis and legs, maintaining this position for as long as possible.
Latissimus Dorsi Muscle Strength Measured by Hand-Held Dynamometer Latissimus Dorsi Muscle Strength Measured by Hand-Held Dynamometer | baseline (week 0) and at the end of intervention (week 8)
  Latissimus dorsi muscle strength will be assessed using a hand-held dynamometer. Participants will be instructed to perform a manual muscle contraction while the dynamometer is placed on the posterior surface of distal humerus. resistance was applied in the direction of shoulder flexion. The maximal force generated during the contraction will be recorded in newtons (N).
Gluteus Maximus Muscle Strength Measured by Hand-Held Dynamometer | baseline (week 0) and at the end of intervention (week 8)
  Gluteus maximus muscle strength will be assessed using a hand-held dynamometer. Participants will be asked to perform a hip extension against the dynamometer placed 5 c m proximal to the knee joint. The maximal force exerted during the movement will be recorded in newtons (N) to assess muscle strength.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy, Cairo Universi, Cairo
  - Faculty of Physical Therapy, Cairo Universi, Giza

REFERENCES:
- [Result] Cashin AG, Booth J, McAuley JH, Jones MD, Hubscher M, Traeger AC, Fried K, Moseley GL. Making exercise count: Considerations for the role of exercise in back pain treatment. Musculoskeletal Care. 2022 Jun;20(2):259-270. doi: 10.1002/msc.1597. Epub 2021 Oct 21. PMID 34676659
- [Result] Calatayud J, Guzman-Gonzalez B, Andersen LL, Cruz-Montecinos C, Morell MT, Roldan R, Ezzatvar Y, Casana J. Effectiveness of a Group-Based Progressive Strength Training in Primary Care to Improve the Recurrence of Low Back Pain Exacerbations and Function: A Randomised Trial. Int J Environ Res Public Health. 2020 Nov 11;17(22):8326. doi: 10.3390/ijerph17228326. PMID 33187076
- [Result] Frizziero A, Pellizzon G, Vittadini F, Bigliardi D, Costantino C. Efficacy of Core Stability in Non-Specific Chronic Low Back Pain. J Funct Morphol Kinesiol. 2021 Apr 22;6(2):37. doi: 10.3390/jfmk6020037. PMID 33922389
- [Result] Wewege MA, Booth J, Parmenter BJ. Aerobic vs. resistance exercise for chronic non-specific low back pain: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2018;31(5):889-899. doi: 10.3233/BMR-170920. PMID 29889056
- [Result] Lorenz D, Morrison S. CURRENT CONCEPTS IN PERIODIZATION OF STRENGTH AND CONDITIONING FOR THE SPORTS PHYSICAL THERAPIST. Int J Sports Phys Ther. 2015 Nov;10(6):734-47. PMID 26618056
- [Result] Tjosvoll SO, Mork PJ, Iversen VM, Rise MB, Fimland MS. Periodized resistance training for persistent non-specific low back pain: a mixed methods feasibility study. BMC Sports Sci Med Rehabil. 2020 May 8;12:30. doi: 10.1186/s13102-020-00181-0. eCollection 2020. PMID 32411374